CLINICAL TRIAL: NCT04423796
Title: Robotic Assisted Early Mobilization in Ventilated ICU Patients: an Interventional Randomized, Controlled Feasibility Study
Brief Title: Robotic Assisted Early Mobilization in Ventilated ICU Patients
Acronym: ROBEM-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Reactive Robotics GmbH (Unknown)
Responsible Party: Principal Investigator, Stefan J Schaller, Deputy Clinical Director, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROBEM I
Record Dates: First submitted 2020-06-06; First posted 2020-06-09 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Critical Illness Polyneuromyopathy; Critical Illness; Early Ambulation; Rehabilitation
Keywords: Early mobilization; pilot trial; feasibility trial; robotic assisted
MeSH Terms: conditions — Critical Illness | interventions — Early Ambulation

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, parallel-group, open label pilot trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic assisted early mobilization (Experimental): Robotic assisted early mobilization started within 72 hours of ICU admission.
  Interventions: Device: Robotic-assisted early mobilization
- Early mobilization (Active Comparator): Early mobilization started within 72 hours of ICU admission without the use of a robotic assistance. Mobilization is done by personell.
  Interventions: Other: Early mobilization

INTERVENTIONS:
Device: Robotic-assisted early mobilization — The early mobilization is done by robotic assistance devices.
  Arms: Robotic assisted early mobilization
Other: Early mobilization — Early mobilization by health care professionals without robotic assistance.
  Arms: Early mobilization

SUMMARY:
Feasibility trial investigating robotic assisted early mobilization vs. early mobilization in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Invasive mechanically ventilated and expected to be ventilated for another 24 hours
* Cardiovascular stability, allowing mobilization
* Respiratory stability, allowing mobilization

Exclusion Criteria:

* Bed-bound before ICU admission
* Bed-rest order or contraindication of weight load of the lower extremity or spine
* Severe skin lesions or fasciitis in the area of contact with the device or rhabdomyolysis
* Fresh SAB, ICB or elevated ICP
* Status epilepticus
* Acute intoxication
* Shock with catecholamine doses >0.3µg/kg/min or acute bleeding including organ ruptures
* Multiorgan failure with lactate > 4 mmol/l
* Body height outside the range 150-195 cm
* Body weight outside the range 45-135 kg
* pAVK IV°
* Pacemakers or other electrical stimulators
* Implanted medical pumps
* Pregnancy
* Life expectancy below 7 days or acute palliative care situation
* Death inevitable or maximum therapy is not carried out by the treating physicians or due to patient's request
* Unable to understand the official language
* ICU stay > 72h at the time of enrolment

Translated with www.DeepL.com/Translator (free version)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2022-08-14 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of early mobilization | Up to Day 5
  Frequency of early mobilization performed by one health care provider during mechanical ventilation

SECONDARY OUTCOMES:
Mobilization level | up to Day 5
  Mobilization level during mechanical ventilation using the ICU Mobility Scale (IMS) ranging from 0-10
Mobilization duration | up to Day 5
  Duration of mobilzation sessions during mechanical ventilation
Frequency of mobilization | up to Day 5
  Frequency of early mobilization during mechanical ventilation
Pain level | up to Day 5
  Pain level at mobilization using a numerical scale (NRS 0-10) or BPS 3-12
Anxiety | up to Day 5
  Anxiety due to mobilization using a numerical scale (NRS 0-10)
Patient satisfaction with mobilization | Up to Day 5
  Satisfaction with mobilization using a numerical scale (NRS 0-10)
Inflammatory response | Up to Day 5
  Zytokin change from before to after mobilization
Health care provider assessment | Up to Day 5
  Assessment of the satisfaction with the mobilization by the health care provider using Likert-Scales (1-5)
Muscle wasting | Up to Day5
  Muscle wasting will be assessed using ultrasound measurement of the M. femoris
Oxygen consumption during mobilization | Up to Day 5
  Oxygen consupmtion during mobilization will be measured using calorimetrie during mobilization
Oesophageal pressure | Up to Day 5
  Oesophageal pressure will be measured during mobilization
Safety events | Up to Day 5
  Frequency of safety events during mobilization

CONTACTS AND LOCATIONS:
Overall Officials: Stefan J Schaller, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Univiversitätsmedizin Berlin, Mitte, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data can be requested from the PI after publication of the study for scientific purpose.
Time Frame: After publishing results.
Access Criteria: Data will be shared to other researchers on reasonable request.

REFERENCES:
- [Derived] Lorenz M, Langer N, Kloss P, Maechler M, Bald A, Warner L, Fuest K, Weiss B, Schaller SJ. ROBotic-assisted Early Mobilization in ventilated surgical critically ill patients (ROBEM-I)-A randomized, controlled, outcome-assessor-blinded pilot study. Anaesth Crit Care Pain Med. 2025 Aug;44(4):101549. doi: 10.1016/j.accpm.2025.101549. Epub 2025 May 23. PMID 40414562